CLINICAL TRIAL: NCT02786849
Title: Neuromuscular Electrical Stimulation During Hemodialysis in Peripheral Muscle Strength and Exercise Capacity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Ana Karla Vieira Brüggemann, Principal Investigator, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1175-1064
Record Dates: First submitted 2016-05-05; First posted 2016-06-01 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Kidney Diseases; Chronic Kidney Diseases; Chronic Kidney Insufficiency; Chronic Renal Insufficiency; Chronic Renal Diseases; Renal Dialysis; Hemodialysis
Keywords: Electric Stimulation; Electric Stimulation Therapy
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Group of high frequency and intensity (Experimental): Group realized high frequency and intensity neuromuscular electrical stimulation
  Interventions: Other: neuromuscular electrical stimulation of high frequency and intensity
- Group of low frequency and intensity (Experimental): Group realized neuromuscular electrical stimulation of low frequency and intensity
  Interventions: Other: neuromuscular electrical stimulation of low frequency and intensity

INTERVENTIONS:
Other: neuromuscular electrical stimulation of high frequency and intensity — Training with neuromuscular electrical stimulation isometric form in lateral and medial bilaterally vast, three times a week, lasting an hour, the first two hours of dialysis.
  Will be applied using portable stimulators with 4 channels. The parameters are: frequency of 50 Hz, pulse width 400ms, rise time and 2s descent, stimulus mode on-off starting with a ratio of 1: 2 in the first week (stimulus time of 10 seconds and rest time of 20s, aiming at adaptation and mitigation of the effects of muscle fatigue), evolving from the second week to a ratio of 1:1 (stimulation time of 10 seconds and rest time of 10s).
  The current intensity is adjusted individually for the first application and gradually increased as the tolerance of patients.
  In each session there will be a warm-up period, training and slowdown. The intensity will be the maximum tolerated by the patient in order increments every session, this being monitored for further evolutionary calculating.
  Arms: Group of high frequency and intensity
Other: neuromuscular electrical stimulation of low frequency and intensity — Training with neuromuscular electrical stimulation isometric form in lateral and medial bilaterally vast, three times a week, lasting an hour, the first two hours of dialysis.
  Will be applied using portable stimulators with 4 channels. The parameters are: 5 Hz frequency, time on: off 1: 3 with a pulse duration of 100ms.
  The current intensity is adjusted individually for the first application and it was the least noticeable by the patient.
  In each session there will be a warm-up period, training and slowdown.
  Arms: Group of low frequency and intensity

SUMMARY:
The objective of this study will be to evaluate the effects of neuromuscular electrical stimulation of high and low frequency and intensity, performed during hemodialysis (HD), on peripheral muscle strength, exercise capacity and muscle change and inflammation markers in patients with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
Clinical trial, randomized, parallel, open, two-arm, blinded assessor, prospective.

Patients with chronic kidney disease on hemodialysis, divided equally into two groups: group of high frequency and intensity neuromuscular electrical stimulation (HG) and a group of low frequency and intensity neuromuscular electrical stimulation (LG).

Randomization was stratified according to gender using 4 block. Drug treatment established for both groups remained unchanged throughout the study period.

Assessments were made on the first working day after hemodialysis, following notification and consent of the medical teams. Patients initially underwent anthropometric measurements and vital signs, later carried out the assessment of peripheral muscle strength, pulmonary function test, submaximal exercise capacity and quality of life questionnaire and depression. After these procedures, the patients were randomized to select HG or LG by opaque envelopes. These evaluations were performed at baseline and after 12 sessions of completion of the protocol.

Furthermore, it was asked to chronic kidney disease (CKD) patients on hemodialysis who presented their latest blood tests clearance index (Kt / V), creatinine, glomerular filtration rate. The evaluation of pro-inflammatory cytokines and regulatory plasma, the enzyme markers of muscle tropism, oxidative stress and muscle injury in patients with CKD was always held at the end of each month as routine clinical.

Two groups conducted training with peripheral electrical stimulation isometric form in lateral and medial bilaterally vast, held three times a week, lasting an hour, the first two hours of dialysis.

Will be applied using portable stimulators with 4 channels. The parameters are:

* HG: frequency of 50 Hertz (Hz), pulse width of 400 microseconds (μs), rise time and fall time of 2 seconds (s), on:off stimulation, initially with a 1:2 relation in the first week (10s of stimulation and 20s of rest, with the objective to adapt and minimize the effects of muscular fatigue), to be increased to a 1:1 relation in the second week (10s of stimulation of and 10s of rest).
* LG: frequency of 5 Hz, on:off stimulation time of 1:3 (10s of stimulation and 30s of rest) with pulse duration of 100 μs.

For both groups, the current intensity was adjusted individually in the first application. In HG, the intensity was gradually increased until visible muscle contraction could be observed: this was the maximum intensity tolerated by the patient. In LG, the intensity was the least noticeable by the patient. These values were monitored for further calculation of intensity evolution throughout the training program.

The blood pressure (BP) will be measured at baseline, and 30 minutes after the end of the session and heart rate (HR) will be monitored every 10 minutes using an oximeter.

In each session there will be a warm-up period, training and slowdown. The first minute will starting with 20% of the intensity value used in the last session with a gradual increase of 20% per minute until 5 minutes, followed by a 50 minute training period and finishing with a 5 minute recovery period gradual reduction of 20% intensity every minute.

Before and after training, patients will be asked about their feelings of fatigue / tiredness of the lower limbs using the modified Borg scale. If reporting muscle pain, the intensity will be assessed by visual analogue scale visual analogue scale (VAS).

They are recruited 76 patients of both sexes, accepted for hemodialysis treatment for at least 6 months. 38 patients are allocated for the HG and 38 to LG.

The sample size calculation was performed in order to advance in GPower 3.1 program based on the results obtained in the study conducted neuromuscular electrical stimulation during hemodialysis in patients with chronic kidney disease. the values of peripheral muscle strength were used before and after treatment respectively 185.4 ± 53 and 222.4 ± 36.6 and the values for the assessment of pre exercise capacity (401.3 ± 55) and post (428.9 ± 69.2) waiting for electrostimulation observe a similar effect. Using an error of 5% (80% test power), it was determined the need for inclusion of 12 patients for the variable peripheral muscle strength and 34 patients for exercise capacity. Recital 10% loss would require the evaluation and treatment of 14 and 38 patients to check the effect on peripheral muscle strength and on exercise capacity respectively.

Safety:

The main negative effect of electrical stimulation is muscle discomfort and / or fatigue of the lower limbs during and after training. Patients will be were asked at the beginning and end of the training on their sense of fatigue / tiredness members, as well as on the feeling of muscle pain. In addition, the current was adjusted individually and gradually increased shape with patient consent. In the case that patients feel a discomfort, the intensity of electric current was reduced, and if required the protocol was stopped by improvement of symptoms.

Statistical analysis:

The data were systematized in IBM SPSS (Statistical Package for Social Sciences) version 20.0. The data were presented as mean ± standard deviation or median and interquartile range and frequency. To verify the data normality the Shapiro-Wilk test was applied. To compare the behavior of the variables between groups was used independent t test for parametric variables and test U Mann Whitney for nonparametric. As for comparing the average pre and post use of electrical stimulation was used ANOVA test for repeated measurements or Friedman test and to check if there is a relationship between respiratory muscle strength and exercise capacity was used Pearson correlation coefficient or Spearman, according to the normal distribution of data. The significance level for the statistical treatment was 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD diagnostic who are on dialysis regularly for at least 6 months, stable and under medical supervision.
* Patients without uncontrolled hypertension, recent ischemic heart disease (3 months or less), unstable angina and severe cardiac arrhythmias.
* Patients without diseases that limit the electrical stimulation protocol (respiratory, orthopedic and / or neurological).
* Patients who do not do any form of physical training or who have been held for more than six months.

Exclusion Criteria:

* Inability to perform any of the study assessments (lack of understanding or collaboration).
* Recent decompensation of the clinical picture with or without hospitalization.
* Presence of chronic obstructive pulmonary disease (COPD or emphysema), musculoskeletal diseases that impede the realization of assessments and training protocol.
* Uncontrolled hypertension, recent ischemic heart disease (3 months or less), unstable angina and severe cardiac arrhythmias.
* Abnormal sensitivity in the lower limbs.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Peripheral muscle strength | one month
  Increased quadriceps strength evaluated by the Isokinetic Biodex System 4 Pro in isometric mode. The highest peak extensor torque is recorded.
Six-minute walk test | one month
  It will be used to evaluate submaximal exercise capacity and will be held in accordance with the recommendations of the American Thoracic Society (Holland et al, 2014.). The larger distance between the two tests will be used for the analysis, this being compared to pre and after training. The reference values are those described by Britto et al., 2013 and an increase of 25 meters after the training will be considered a clinically important improvement.

SECONDARY OUTCOMES:
Pulmonary function test | one month
  performed with the portable digital spirometer the following parameters are obtained with the same maneuver: forced vital capacity (FVC) in liter, forced expiratory volume in one second (FEV1) in liter and the FEV1/FVC ratio expressed in absolute terms and in percentage of predicted values normality according to the determined by Pereira et al. (2007).
Quality of life | one month
  It will be measured using the questionnaire Kidney Disease and Quality-of-Life Short Form (KDQOL-SF), the degree of commitment of each domain is measured by values ranging from zero (greater degree of commitment) 100 (no impairment). Thus, the higher the score, the better the quality of life. The questionnaire will be pre to post intervention to see if there were improvements.
Anxiety and Depression | one month
  It used the Hospital Anxiety and Depression Scale - HADS (Hospital Anxiety and Depression Scale). The overall scores for each subscales (anxiety or depression) ranges from 0 to 21, where 0 corresponds to the lowest level of depression or anxiety and 21 at most. At the end, add up the scores of anxiety and depression. The scale is reapplied to the end of the training to compare the scores.
urea clearance | one month
  The result of the urea clearance rate is obtained by multiplying the clearance of the dialyzer (clearance, K, in mL / min) by the planned dialysis time (t in min), and divide the result by the volume of distribution of the patient solute ( volume in ml, for the urea this corresponds to 60% of patient weight).
glomerular filtration rate | one month
  The result of glomerular filtration rate is obtained by NefroCalc calculation system, selecting the CKD-EPI function that is based on the amount of creatinine in mg / dL, age, gender, and individual class, generating the value of the filtration rate glomerular in mL / min / 1.73m2.
pro and anti-inflammatory cytokines | one month
  Both pro and anti-inflammatory cytokines will be analyzed using the plasma of patients with CKD during hemodialysis. Samples of 4 ml of blood will be taken from existing fistulas in patients, there is no need, therefore, no additional invasive procedure for collection. The assessment using the method of enzyme-linked immunosorbent assay (ELISA) using a kit suitable for this purpose.
muscle trophism markers | one month
  The muscle trophism markers will be analyzed using the plasma of patients with CKD during HD. Samples of 4 ml of blood will be taken from existing fistulas in patients, there is no need, therefore, no additional invasive procedure for collection. The assessment of changes in markers related to muscle tropism (mTOR and BDNF - Brain derivated neurotrophic factor) will be evaluated by Western blot.
oxidative stress | one month
  Samples of approximately 200 uL plasma will be reserved for analysis of the total glutathione (GSH) levels. Glutathione is measured by the method Tieze.
markers of muscle damage | one month
  After the coagulated blood samples are centrifuged for serum separation, despising the figurative elements and avoiding hemolysis according to the procedures recommended for biochemical analysis. Dosages of CK and LHD will be carried out with the aid of specific reagent kits for each analysis and quantified by spectrophotometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Karla Vieira Brüggemann, Santo Amaro da Imperatriz, SC - Santa Catarina, Brazil

REFERENCES:
- [Derived] Bruggemann AK, Mello CL, Dal Pont T, Hizume Kunzler D, Martins DF, Bobinski F, Pereira Yamaguti W, Paulin E. Effects of Neuromuscular Electrical Stimulation During Hemodialysis on Peripheral Muscle Strength and Exercise Capacity: A Randomized Clinical Trial. Arch Phys Med Rehabil. 2017 May;98(5):822-831.e1. doi: 10.1016/j.apmr.2016.12.009. Epub 2017 Jan 16. PMID 28093194